CLINICAL TRIAL: NCT00590109
Title: Germline BRCA1 and BRCA2 Mutations in Jewish Women Affected by Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sarah Lawrence College (Other); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: 97-029; CA08748
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Jewish; BRCA1; BRCA2; 97-029
MeSH Terms: conditions — Breast Neoplasms | interventions — Hematologic Tests; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Blood test; Other: Questionnaire

INTERVENTIONS:
Other: Blood test — subjects will provide one 8ml blood sample drawn into one ACD tube and 16ml of blood drawn into two EDTA (purple top) tubes.
Other: Questionnaire — A questionnaire encompassing medical, environmental exposure, and reproductive history.

SUMMARY:
The purpose of this project is to further characterize inherited predisposition to breast cancer mediated by specific BRCA alleles (BRACA1 185delAG and 5382insC; BRCA2 6174delT) among Jewish women.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for the study if they are over 18 years of age, identify their ancestry as Jewish (both Sephardic and Ashkenazi Jews are eligible), have or have had a diagnosis of breast cancer, and are able to give informed consent.
* Relatives, age 18 or older, of the patients who meet eligibility criteria above and are found to have a specific BRCA1 or BRCA2 mutation if they are able to give informed consent.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A list of Jewish women diagnosed with breast cancer at Memorial Hospital after January 1994 will be generated from the hospital database. Patients that meet the study criteria will have a letter sent to their oncologist asking permission to invite the patient to participate in a study.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 1997-03; Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
to further characterize inherited predisposition to breast cancer mediated by specific BRCA alleles among Jewish women. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org